CLINICAL TRIAL: NCT03635970
Title: Microvascular Effect After the Application of Cell Therapy With a Hematopoietic Stem Cell Concentrate in Patients With Peripheral Arterial Disease With Non-critical Ischemia and Diabetes
Brief Title: Cell Therapy for Peripheral Arterial Disease and Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Regional de Alta Especialidad del Bajio (Other)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIBIUG-P14-2018
Record Dates: First submitted 2018-07-06; First posted 2018-08-17 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Peripheral Arterial Disease; Diabetes Mellitus
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Treatment for peripheral arterial disease plus diabetes with 2 arms of study.
Who Masked: Outcomes Assessor
Masking Description: the evaluator of the treatment goals does not know the treatment that each patient received
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional treatment (Placebo Comparator): receive the best conventional therapy
  Interventions: Procedure: celular therapy
- experimental treatment (Active Comparator): The best medical treatment possible plus celular therapy
  Interventions: Procedure: celular therapy

INTERVENTIONS:
Procedure: celular therapy — application of cell therapy with a concentrate of hematopoietic progenitor cells or celular therapy

SUMMARY:
This is a randomized controlled trial with blinding (for the observer who evaluates treatment goals).

With two groups to study. A group of patients with conventional therapy for the treatment of PAD (Platelet antiaggregant, statin, cilostazol in case of claudication) and the other group of patients with conventional therapy for treatment of PAD plus cell therapy with objective to evaluate the microvascular effect after the application of cell therapy with a hematopoietic stem cell concentrate in patients with PAD with non-critical ischemia and Diabetes. Perform evaluations of the microcirculation by means of TcPO2 at 30, 60, 90 and 180 days after the experimental maneuver (cell therapy) and conventional therapy.

DETAILED DESCRIPTION:
INTRODUCTION: Peripheral arterial disease (PAD) is defined as arterial occlusion of the lower extremities. Based on epidemiological studies using the Ankle-Brachial Index (ABI), the prevalence of PAD (defined as an ABI <0.9) in diabetic patients ranges from 20% to 30%. Diabetic patients with PAD have a higher mortality and death rate at a younger age than patients without diabetes. The appropriate medical treatment for EAP in patients with diabetes is based on the control of cardiovascular risk factors. Revascularization is indicated in particular situations in PAD in the context of critical chronic ischemia (ABI <0.6), however, anatomical factors, operative risk, technical difficulties or patient preferences may limit its use in patients with PAD and diabetes. Therapeutic angiogenesis is an experimental approach to restore perfusion and cell therapy can provide a continuous source of growth factors and structural elements for therapeutic angiogenesis. The transcutaneous oxygen pressure (TcPO2) is defined as a microvascular evaluation system. The microvascular effect of cell therapy at an earlier stage of PAD has not been analyzed as non-critical ischemia in patients with diabetes.

OBJECTIVE: To evaluate the microvascular effect after the application of cell therapy with a concentrate of hematopoietic stem cell in patients with PAD with non-critical ischemia and Diabetes.

MATERIAL AND METHODS: Randomized controlled clinical trial with blinding (for the observer who evaluates treatment goals). With two groups for your study. A group of patients with conventional therapy for the treatment of PAD (Platelet antiaggregant, statin, cilostazol in case of claudication) and the other group of patients with conventional therapy for treatment of PAD plus cell therapy, to be carried out in patients entitled to the Mexican Institute of the Social Security of the Guanajuato Delegation, with diagnosis of Diabetes Mellitus type 2 of more than 10 years of detection and with diagnosis of peripheral arterial disease with an ABI between 0.6 and 0.9 that agree to participate in the study. Cell therapy will consist of hematopoietic progenitor cells identified as a fraction of cells identified by flow cytometry as CD34 + obtained by peripheral blood harvesting procedure, prior mobilization process with filgrastim.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with affiliation to the Mexican Institute of Social Security.
2. Patients older than 35 years.
3. Patients with Type 2 Diabetes Mellitus over 10 years of detection.
4. Patients with Peripheral Arterial Disease with ABI between 0.6 and 0.9.
5. Signature of informed consent.

Exclusion Criteria:

1. Patients with a history of uncontrolled oncological disease in the last 5 years.
2. Presence of Chronic Renal Insufficiency with a calculated creatinine clearance using a Cockcroft formula less than 15ml / min.
3. Ulcer that defines diabetic foot or tissue necrosis that requires partial or total amputation of a limb.
4. Serious active infectious process anywhere in the body.
5. Have restrictions with the use of filgrastim such as treatment with lithium, chemotherapy or radiotherapy, as well as a history of autoimmune thrombocytopenia, vasculitis, previous cardiovascular disease, Sweet's syndrome or Steven-Johnson syndrome.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
TcPO2 | 180 days
  Change is being assessed, through the transcutaneous pressure of oxygen, after the application of the therapies

CONTACTS AND LOCATIONS:
Overall Officials: B MURILLO, MD, Study Director — IMSS
Locations (1):
- Instituto Mexicano Del Seguro Social, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Via email, the researchers can request information about study
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available in every time and after one year after its publication
Access Criteria: Via email, the researchers can request information about study